CLINICAL TRIAL: NCT03262480
Title: Perioperative Goal Directed Fluid Therapy During Radical Cystectomy: the Impact of Stroke Volume Optimization vs Dynamic Central Venous Pressure
Brief Title: The Stroke Volume Optimization of Goal Directed Fluid Therapy During Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Mahmoud Othman, professor of Anesthesia and surgical ICU, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MD/17.07.27
Record Dates: First submitted 2017-08-14; First posted 2017-08-25 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Radical Cystectomy

STUDY DESIGN:
Intervention Model Description: Two groups:
  * Stroke volume optimization group (SVO group).
  * Central venous pressure dynamic group(CVPdyngroup).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The management will be carried out by a member of research team only aware of allocation group. The attending anesthesiologist, surgeons and nursing staff will be totally blind of randomization schedule or the hydration regimen used. All postoperative clinical staff handling patient care will be also unaware of the aim of the work.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke volume optimization (Active Comparator): Colloid aliquots of 200 ml 6% hydroxy ethyl starch 130/ 0.4 (Voluven) will be administered within 10 minutes and stroke volume response will be recorded .If stroke volume increase by more than 10 % for 20 minutes, the aliquot will be repeated.
  Interventions: Other: stroke volume optimization
- Central venous pressure dynamic (Sham Comparator): Colloid aliquots of 200 ml 6% hydroxy ethyl starch 130/ 0.4(Voluven) will be administered within 10 minutes and CVP response will be recorded. If CVP failed to rise sustainably for more than 2 mmHg for 20 minutes, the aliquot will be repeated.
  Interventions: Other: stroke volume optimization

INTERVENTIONS:
Other: stroke volume optimization — Hemodynamic variables including stroke volume (SV), stroke volume variation (SVV), stroke volume index (SVI), cardiac output (COP), cardiac index (CI), systemic vascular resistance (SVR), systemic vascular resistance index (SVRI), thoracic fluid content (TFC), corrected flow time (FTC), index of contractility (ICON), systolic time ratio (STR), oxygen delivery (DO2) and oxygen delivery index (DO2I) will be measured by Cardiac output non-invasive monitor (ICONTM, OSYPKA medical cardiotronic GMBH, Elixir, Germany). Heart rate (HR), mean arterial blood pressure (MAP), central venous pressure (CVP) and arterial oxygen saturation (Sao2) will be measured using HP monitor.
  If mean arterial blood pressure(MAP) drops below 65 mmHg despite achievement of SVopt and CVPmax in both groups, a bolus dose of 5 mg ephedrine will be given and repeated as needed .Norepinephrine will be given for persistent hypotension.Dobutamine 5 mic/kg/min will be started if cardiac index less than 2.5 l/m2.
  Other Names: central venous pressure dynamic

SUMMARY:
Although fluid therapy is of paramount value in anesthetic practice, there is no guideline available for perioperative fluid management in major abdominal surgery. So, there is a need to establish whether goal directed fluid therapy protocol is effective during radical cystectomy and urinary diversion. A balance of perioperative fluid therapy is crucial, yet the method to achieve this equilibrium remains a highly debated subject. Therefore, this study will be designed to investigate the effects of two individualized goal directed fluid therapy during radical cystectomy to encourage an effective circulating blood volume and pressure. Accordingly, as a primary outcome, the investigators assume that stroke volume optimization could maintain better perioperative hemodynamic stability with low incidence and severity of hypotensive episodes together with achievement of maximal oxygenation. Hopefully this regimen could help to decrease the possibility of perioperative tissue hypoperfusion and the possible associated complications as a secondary outcome.

DETAILED DESCRIPTION:
Study protocol:

Patients will be randomly assigned to one of two equal groups, according to computer-generated randomization sequence into:

* Stroke volume optimization group (SVO group).
* Central venous pressure dynamic group(CVPdyngroup).

Stroke volume optimization group (SVO group):

Colloid aliquots of 200 ml 6% hydroxy ethyl starch 130/ 0.4 (Voluven, Fresenius kabi, Deutschland GmbH, Bad Homburg, Germany) will be administered within 10 minutes and stroke volume response will be recorded .If stroke volume increase by more than 10 % for 20 minutes, the aliquot will be repeated. No further aliquots will be given once stroke volume failed to increase >10%. The last stroke volume without rise of > 10% will be defined as optimum stroke volume (SVopt).When stroke volume decreases by 10% below (SVopt), this will be defined as trigger stroke volume (SVT). Stroke volume will be followed every 30 minutes during surgery and every 4 hours for 24 hours postoperatively .

Central venous pressure dynamic group (CVPdyn group):

Colloid aliquots of 200 ml 6% hydroxy ethyl starch 130/ 0.4(Voluven) will be administered within 10 minutes and CVP response will be recorded. If CVP failed to rise sustainably for more than 2 mmHg for 20 minutes, the aliquot will be repeated. No further aliquots will be given once CVP increases more than 2 mmHg above the recorded one.The last CVP with sustained rise of>2 mmHg will be defined as CVP maximum (CVPmax).When CVP decrease below (CVPmax)by 3 mmHg, this will be defined as trigger CVP (CVPT).CVP will be followed every 30 min during surgery and every 4 hours for 24 hours postoperatively

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with American Society of Anesthesiologists (ASA) physical status I - II scheduled for radical cystectomy and urinary diversion for muscle invasive urinary bladder carcinoma .
* Both sexes

Exclusion Criteria:

* Patients younger than 18 years
* Body mass index (BMI) < 25 and >35.
* Patients with any contraindications to epidural anesthesia (patient refusal, local skin infection, previous spine surgery and coagulopathy).
* Those with known allergy to local anesthetics.
* Patients with major cardiovascular problems with ejection fraction < 40 .
* Renal impairment with serum creatinine >1.8 mg/dl
* Patients with hepatic dysfunction will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Perioperative hypotension | perioperative
  Mean arterial blood pressure < 65mmHg
Maximal tissue oxygenation | perioperative
  Oxygen delivery index > 550 ml/min/m2

SECONDARY OUTCOMES:
Medical postoperative complication | 48 hours postoperative
  Acute kidney injury (AKI) . Postoperative serum creatinine value is either more than 1.5-fold or more than 0.3 mg/dl before surgery within 48 hours
Surgical postoperative complication | 7-days postoperative
  Nausea, vomiting, abdominal distension, anastomotic leakage, paralytic ileus
Anesthetic postoperative complication | 24 hours postoperative
  Cardiogenic pulmonary edema.Cardiac index < 2.5 l/min/m2
Surgical postoperative complication | 7-days postoperative
  Wound infection and burst abdomen
Respiratory postoperative complication | 7-days postoperative
  Pneumonia, acute respiratory distress, postoperative ventilation and ICU admission.length of ICU stay in days.
Postoperative complication | 7-days postoperative
  mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M Othman, Professor, Principal Investigator — Mansoura faculty of medicine
Locations (1):
- Urology and nephrology center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided